CLINICAL TRIAL: NCT01973998
Title: Effects of Roflumilast in Hospitalized COPD on Mortality and Re-hospitalization
Brief Title: Effects of Roflumilast in Hospitalized Chronic Obstructive Pulmonary Disease( COPD) on Mortality and Re-hospitalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Gerard Criner, Chief of Pulmonary and Critical Care Medicine, Temple University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21474
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: COPD
Keywords: COPD; Emphysema; Roflumilast; readmission
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Experimental): 500 ug tablet daily for 180 days
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Placebo 1 tablet daily x 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — PDE4 inhibitor
  Other Names: Daliresp
  Arms: Roflumilast
Drug: Placebo — Inactive substance.
  Other Names: Inactive substance
  Arms: Placebo

SUMMARY:
Background: COPD exacerbations add considerably to patients' burden because they: (1) cause frequent hospital admissions and relapses or readmissions, (2) contribute directly to the death of many patients, either during hospitalization or shortly thereafter, (3) cause patients significant stress, prolonged physical discomfort, disability and dramatically reduced quality of life, (4) consume the majority of the resources available to manage this chronic condition, (5) frequently progress to a severe stage warranting hospitalization before any abortive treatment is instituted, and (6) may hasten the progressive loss of lung function, a steady decline that is a cardinal feature of COPD itself. Hence, investigations of new therapies to treat COPD patients who are hospitalized with a severe exacerbation are desperately needed.

Objective: To test the feasibility of roflumilast to decrease all cause readmission and mortality 180 days after hospitalization for acute COPD exacerbation.

Methods: Parallel-group, prospective, randomized, double blind, placebo-controlled trial of roflumilast 500 ug daily vs. placebo in approximately 100 hospitalized AECOPD patients. Inclusion Criteria. Primary diagnosis of AECOPD; admission to the hospital <12 hours; patient age >40, < 80 years old; cigarette smoking > 10 pack-years. Exclusion Criteria. Prior diagnosis or high suspicion for asthma; pulmonary edema, pneumonia, interstitial lung disease or significant bronchiectasis; intubated and mechanically ventilated at the time of evaluation; active liver disease, or transaminase elevations (> 3xULN); history of heavy ethanol use; history of suicidal behavior ≤ 2 years or suicidal ideation ≤ 6 months prior to enrollment; pregnant or lactating females. Those on the following excluded medications: P450 inducers and CYP3A4 inhibitors or dual inhibitors that inhibit both CYP3A4 and CYP1A2 simultaneously

DETAILED DESCRIPTION:
Background :Chronic obstructive pulmonary disease (COPD) afflicts 24 million US residents and is the 3th leading cause of death in the United States. Each year, 150,000 patients die from COPD in the U.S. or about one patient every 4 minutes. Health care costs for COPD patients in the US is approximately $6.5 billion/ year, but its indirect costs probably double the costs of care when taking into account lost productivity and caretaker expenses. COPD exacerbations add considerably to that burden because they: (1) cause frequent hospital admissions and relapses or readmissions, (2) contribute directly to the death of many patients, either during hospitalization or shortly thereafter, (3) cause patients significant stress, prolonged physical discomfort, disability and dramatically reduced quality of life, (4) consume the majority of the resources available to manage this chronic condition, (5) frequently progress to a severe stage warranting hospitalization before any abortive treatment is instituted, and (6) may hasten the progressive loss of lung function, a steady decline that is a cardinal feature of COPD itself.

Hospitalized exacerbations result in a profound impact on patient survival, function, symptoms and health status as well as costs. Re-hospitalization in COPD is frequent and associated with a particularly negative impact. Patients discharged from the hospital after a COPD exacerbation have a high mortality and are frequently readmitted with recurrent exacerbations. Although a number of pharmacologic and behavioral interventions have been used to decrease exacerbations in COPD, it is not clear that these same interventions are successful in reducing hospital admission rates or re-admission rates. Except for the use of noninvasive ventilation in patients that present in acute respiratory failure during COPD hospitalization, no new therapies have been discovered in the last 3 decades.

A. Specific Aims: In this pilot proposal, we will test the feasibility of roflumilast to decrease all cause readmission and mortality 180 days after hospitalization for acute COPD exacerbation. We propose to conduct this study in 100 patients at three centers to assess the tolerance and treatment effect of roflumilast in order to power an appropriate definitive phase III multicenter trial.

B. Study Design and Synopsis: Parallel-group, prospective, randomized, double blind, placebo-controlled trial of roflumilast 500 ug daily vs. placebo in approximately 100 hospitalized AECOPD patients. Both groups will receive GOLD guideline-recommended care.

Patients hospitalized with AECOPD will be eligible for enrollment ≤ 12 hours after admission. Demographics, blood tests, health related quality of life, comorbidity (Deyo-Charlson index), post bronchodilator spirometry, vital signs, dyspnea measured by MMRC, SaO2 and amount of inspired O2 to maintain SaO2> 90% at rest, serum fibrinogen levels, HBA1c, Biomarkers and Genetics will be obtained after enrollment and then patients will be randomized to standard AECOPD care plus roflumilast 500 ug daily vs. placebo. Patients will begin roflumilast or placebo < 12 hours of hospitalization for a total period of 180 days post enrollment. On discharge day (approximately day 3-4 after admission based on the recent COPD CRN zileuton study of hospitalized AECOPD), the measurements will be repeated as indicated (baseline measurements), with follow-up phone assessments at days 7, 30, 60, 90, 120 and 194 days post enrollment. An in-person clinical visit will be conducted at days 14 and 180 post randomization.

Study will begin within 12 hours of patient's admission and last for 194 days. Baseline: Will occur within 12 hours of patient's admission to the hospital. Patients will have a medical history taken as well as smoking history. Patients will also be given a physical exam including vital signs. A spirometry test will also be performed. Women with the potential to become pregnant will be given a pregnancy test. Data will also be collected in regards to dyspnea scales, Deyo-Charlson index, and GOLD classification. Patients will complete a Columbia Suicide Severity Rating Scale to exclude patients with a history of suicidal behavior ≤ 2 years or suicidal ideation ≤ 6 months prior to enrollment Randomization: Patients will be randomized to one of two treatment groups. Randomization will be done using a randomized block design stratified by treatment center. One group will receive roflumilast 500 mcg (Daliresp®) and the other will receive a placebo tablet. Patients will begin one of these treatment arms within 12 hours of hospitalization for a total period of 180 days post enrollment.

Day of hospital discharge: A spirometry test will be performed and an adverse event assessment will be completed.

Day 7: Phone Visit. Data collected includes: interim history, adverse events, vital status, and exacerbation history. During this telephone visit the study doctor or nurse coordinator will ask how the patient is feeling and if they have needed to visit the doctor or go to the emergency room or hospital since the last time they were contacted. They will be asked how well they are tolerating the study drug.

Day 14: Clinic Visit. At this visit vital signs, C-SSRS test, interim history, adverse event assessment, vital status, and exacerbation history will be recorded. The following questionnaires will given: EQ-5D, the St. George's Respiratory Questionnaire (SGRQ), and the Modified Medical Research Council dyspnea score (MMRC).

Days 30, 60, 90, & 120: Phone Visit. Data to be collected includes: interim history, adverse events assessments, vital status, and exacerbation history. During each of these telephone visits the study doctor or nurse coordinator will ask how the patient is feeling and if they have needed to visit the doctor or go to the emergency room or hospital since the last time they were contacted. They will be asked how well they are tolerating the study drug.

Day 180: Clinic Visit. At this visit vital signs, C-SSRS test, interim history, adverse event assessment, vital status, and exacerbation history will be recorded. A spirometry test will be performed as well during this visit. The following questionnaires will given: EQ-5D, the St. George's Respiratory Questionnaire (SGRQ), and the Modified Medical Research Council dyspnea score (MMRC).

Day 194: Phone Visit. This phone call covers the wash out period for the study treatments. Data to be collected includes: interim history, adverse events assessments, vital status, and exacerbation history. During this telephone visits the study doctor or nurse coordinator will ask how the patient is feeling and if they have needed to visit the doctor or go to the emergency room or hospital since the last time they were contacted.

All patients will receive standardized, optimized care for AECOPD. Nebulized albuterol (2.5 mg in 0.5 ml, dilute to 3 ml NSS administered every 4-6 hours) and ipratropium bromide (0.5 mg in 0.5 ml, diluted with 2.5 ml of saline administered every 6 hours) will be given. A 14-day course of systemic steroids consisting of intravenous methylprednisolone 125 mg every 6 hours for up to 72 hours, followed by once daily oral prednisone 60mg/day for days 4-7, 40 mg prednisone days 8-11 and 20 mg prednisone days 12-14 will be provided. A 7-day course of antibiotics will be selected based on patient's medical allergy history and relevant culture data if available. Supplemental oxygen will be provided by route and dose to achieve maximum patient comfort and compliance to maintain a SaO2 > 92%. Noninvasive positive pressure ventilation will be utilized at the discretion of the treating physicians.

Following oral administration, roflumilast is rapidly absorbed with a tmax of about 1 hour and an 80% bioavailability. Roflumilast is metabolized by CYP3A4 and CYP1A2 enzymes with N-oxide being the principal major metabolite. N-oxide has selectivity for the PDE4 isoenzyme and mainly accounts for roflumilast's in vivo bioactivity. No major interactions have been reported between roflumilast and other COPD medications.

The present proposal is a pilot study designed to test the feasibility of a future project to be conducted in a multicenter trial in hospitalized patients. Determine the treatment effect of roflumilast as add-on therapy to decrease all cause readmission and mortality as a composite endpoint 180 days after randomization to roflumilast or matching placebo ≤ 12 hours after hospitalization for acute COPD exacerbation.

The primary analysis for all study outcomes will be performed on an intention to treat basis. In the intention to treat approach, all subjects are analyzed in the group to which they were randomized, regardless of whether the assigned treatment was adhered to and regardless of whether there were any eligibility violations.

Univariate descriptive statistics will be calculated for baseline parameters overall and by treatment group. For categorical outcomes, these will include the number percentage of subjects in each category. For continuous variables, these will include the mean and standard deviation for variables with approximately normal distributions and the median and 25th and 75% percentiles for variables with skewed distributions.

The primary outcome is time from randomization to a composite outcome of all cause re-hospitalization and all-cause mortality, whichever comes first. The primary analysis will be a log-ranked test and associated Kaplan-Meier plot, unadjusted for any covariates. Censoring will occur at the earliest date of any of the following occurrences, unless the subject has already experienced the primary outcome event:

* Lost to follow-up despite intensive efforts
* Subject or healthcare proxy withdrawal of consent
* 180 days after randomization. 3. Analysis of secondary outcomes. Primary analysis of other time to event outcomes will be performed using unadjusted log rank tests that have associated Kaplan-Meier plots, similar to the primary analysis of the primary study outcome. Secondary analysis of these outcomes will use Cox regression to adjust for baseline subject factors (covariates) that are known to be associated with the outcome.

The primary analyses of changes in continuous measures such as absolute and percent changes in spirometry and dyspnea scores, for example, will be analyzed using an analysis of covariance where change from baseline to a particular time period is the dependent variable.

In this pilot proposal, the treatment effect of roflumilast vs. placebo to prolong the time to event of a combined endpoint of death or re-hospitalization will be assessed in an intention to treat manner. In a similar manner, the treatment effect of roflumilast vs. placebo to effect all of the secondary endpoints proposed to be measured in the pivotal phase III trial will also be measured (time to respiratory death or respiratory re-hospitalization during the 180 days post-randomization; rate of death or readmission at 30 days post-discharge; treatment failure; change in health status, change in FEV1, and dyspnea during the 180 days post-randomization; length of hospital stay during the index hospitalization; and the tolerance of roflumilast vs. placebo in hospitalized AECOPD).

Because this is a pilot study the intent is to see if there is a signal that would justify a larger clinical trial. Therefore the significance level has been set to 0.1 and the power has been set at 0.7. A total of 100 patients will enter this two treatment parallel-design study. The probability is 70 percent that the study will detect a treatment difference at a two sided 10.0 percent significance level, if the true hazard ratio is 1.654. This is based on the assumption that the accrual period will be 36 months and the follow up period will be 6 months and the median time to event is 8 months. The total number of events will be 73.

ELIGIBILITY:
Inclusion Criteria:

Primary diagnosis of AECOPD defined as acute increase in dyspnea, sputum volume, and/or sputum purulence without other identified cause; admission to the hospital <12 hours; patient age >40, < 80 years old; cigarette smoking > 10 pack-years; informed written consent.

Exclusion Criteria:

Prior diagnosis or high suspicion for asthma based on investigator judgment; pulmonary edema, pneumonia, interstitial lung disease or significant bronchiectasis based on admission chest x-ray; intubated and mechanically ventilated at the time of evaluation; active liver disease, or transaminase elevations (> 3xULN); history of alcoholism or heavy ethanol use; history of suicidal behavior ≤ 2 years or suicidal ideation ≤ 6 months prior to enrollment; pregnant or lactating females. Those on the following excluded medications: P450 inducers (e.g., rifampicin, phenobarbital, carbamazepine, and phenytoin) and CYP3A4 inhibitors or dual inhibitors that inhibit both CYP3A4 and CYP1A2 simultaneously (e.g., erythromycin, ketoconazole, fluvoxamine, enoxacin, cimetidine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-11; Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Criner, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data will be in a de-identified computerized dataset maintained by the investigators at Temple University. De-identified data will be shared through either password protected website maintained without cost to researchers after requests are vetted by principal investigators at Temple University.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal as determined by the investigators at Temple University.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 33 | 35
Completed | 31 | 33
Not Completed | 2 | 2
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7) | 59.3 (8.1) | 59.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 21 | 41
  White | 2 | 3 | 5
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Time to All-cause Mortality or Re-hospitalization During the 180 Days Post-randomization.
Description: A combined endpoint of time to all-cause mortality or re-hospitalization during the 180 days post-randomization was used.
Time Frame: 180 days
Population: Patients who completed 180 days of follow-up
Measure: Mean (80% Confidence Interval); unit: Days to event
Units Other Than Participants: Number of hospitalizations
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 31 | 33
Number analyzed (Number of hospitalizations) | 21 | 29
Days to event | 54 [41.9 to 66.1] | 55 [43.6 to 66.4]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Equivalence — The primary outcome is time from randomization to a composite outcome of all cause re-hospitalization and all-cause mortality, whichever comes first. The primary analysis will be a log-ranked test and associated Kaplan-Meier plot, unadjusted for any covariates; p < 0.1, Log Rank — Because this is a pilot study the intent is to see if there is a signal that would justify a larger clinical trial. Therefore the significance level has been set to 0.1 and the power has been set at 0.7; Hazard Ratio (HR) = 1.654, 10% CI 2-sided [1.175 to 2.133], Standard Deviation .4789
Statistical Analysis 2: Comparison: Roflumilast vs Placebo; A total of 100 patients is required in a 2 treatment parallel-design study. There is a 70% probability that the study will detect a treatment difference at a 2-sided 10% significance level, if the true hazard ratio is 1.654. This is based on the assumption that the accrual period will be 36 months and the follow up period will be 6 months and the median time to event is 8 months. The total number of events will be 73; Test type: Superiority; p = 0.1, Log Rank; Hazard Ratio (HR) = 1.654, 10% CI 2-sided [1.175 to 2.133], Standard Deviation .4789

2. Secondary Outcome: Respiratory Death or Respiratory Re-hospitalization
Description: respiratory death or respiratory re-hospitalization during the 180 days post-randomization; rate of death or readmission during the 30 days post-discharge; treatment failure (see definition below); change in health status, FEV1 (forced expiratory volume at one second, and dyspnea during the 180 days post-randomization; length of hospital stay during the index hospitalization.
Time Frame: 180 days
Measure: Number; unit: number of events
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 31 | 33
number of events | 21 | 29

3. Other Pre Specified Outcome: Assess Tolerance of Roflumilast vs. Placebo in Hospitalized AECOPD
Description: Reported adverse events during the course of the study. Need to withdraw study drug due to adverse events
Time Frame: 180 days
Measure: Number; unit: reported events
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 31 | 33
reported events
  Diarrhea | 8 | 10
  Weight loss | 7 | 3
  Nausea | 11 | 4
  Headache | 12 | 15
  Back pain | 13 | 16
  Insomnia | 16 | 15
  Decreased appetite | 10 | 8
  Dizziness | 9 | 8
  Depression | 8 | 8

ADVERSE EVENTS:
Time Frame: 180 days
Description: Death was not considered an adverse event as it was part of the combined study endpoint
Arm/Group | Roflumilast | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 13/31 | 16/33
Other Adverse Events (participants affected / at risk) | 16/31 | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=31) | Placebo (N=33)
Rehospitalization (Respiratory, thoracic and mediastinal disorders) | 13 (31) | 16 (35)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=31) | Placebo (N=33)
diarrhea (Gastrointestinal disorders) | 8 (8) | 10 (10)
Weight loss (General disorders) | 7 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 11 (11) | 4 (4)
Headache (Nervous system disorders) | 12 (12) | 15 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 16 (16)
Insomnia (Nervous system disorders) | 16 (16) | 16 (16)
Decreased appetite (Gastrointestinal disorders) | 10 (10) | 8 (8)
Dizziness (Nervous system disorders) | 9 (9) | 8 (8)
Depression (Nervous system disorders) | 8 (8) | 8 (8)

LIMITATIONS AND CAVEATS:
Small sample size, short duration of exposure (6 months), single center nature, absence of chronic bronchitic symptoms in all subjects and lack of mortality events as a measurable endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT01973998/Prot_SAP_000.pdf